CLINICAL TRIAL: NCT03602053
Title: An Open-label, Randomized, Controlled, Single Centre, Phase IIb Study to Assess the Immunogenicity, Reactogenicity and Safety of Three Live Oral Rotavirus Vaccines, ROTAVAC® , ROTAVAC 5CM and Rotarix® in Healthy Zambian Infants
Brief Title: Study of BBIL's ROTAVAC® and ROTAVAC 5CM Vaccines in Zambia
Acronym: ROTAVAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: PATH (Other); Christian Medical College, Vellore, India (Other); Children's Hospital Medical Center, Cincinnati (Other); Bharat Biotech International Limited (Industry)
Responsible Party: Principal Investigator, Roma Chilengi, Chief Scientific Officer, Centre for Infectious Disease Research in Zambia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVIA 066
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Diarrhea; Diarrhea Rotavirus
Keywords: diarrhea; Rotavirus; ROTAVAC; Rotavirus vaccine
MeSH Terms: conditions — Diarrhea | interventions — RIX4414 vaccine

STUDY DESIGN:
Intervention Model Description: Phase IIb, single center, randomized, controlled, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ROTAVAC 5D (Experimental): Bharat Biotech International Ltd's new Rotavirus vaccine, ROTAVAC 5D is a live, attenuated G9P[11] monovalent vaccine at a dose of 0.5mL containing NLT log 10^5.0 focus forming units (FFU) per dose. 5D is in liquid form.
  Interventions: Biological: ROTAVAC 5D
- ROTAVAC® (Experimental): Bharat Biotech International Ltd's licensed rotavirus vaccine, ROTAVAC® is a live, attenuated G9P[11] monovalent vaccine at a dose of 0.5mL containing NLT log 10^5.0 focus forming units (FFU) per dose. ROTAVAC® is in frozen form and is thawed till fully liquid prior to administration.
  Interventions: Biological: ROTAVAC®
- Rotarix® (Active Comparator): GSK Biologicals' licensed rotavirus vaccine, Rotarix® is a live attenuated RIX4414 strain of human rotavirus of the G1P[8] type containing not less than 106.0 CCID50 (cell culture infectious dose 50%) of the RIX 4414 strain of human rotavirus.
  Interventions: Biological: Rotarix®

INTERVENTIONS:
Biological: ROTAVAC® — 0.5 ml of the vaccine will be administered orally thrice at 6, 10 and 14 weeks of age.
  Arms: ROTAVAC®
Biological: ROTAVAC 5D — 0.5 ml of the vaccine will be administered orally thrice at 6, 10 and 14 weeks of age.
  Arms: ROTAVAC 5D
Biological: Rotarix® — 1.5 ml of the liquid vaccine will be administered orally twice at 6 and 10 weeks of age.
  Arms: Rotarix®

SUMMARY:
The study is being conducted to evaluate and compare the immunogenicity of ROTAVAC® and ROTAVAC 5D 28 days after the last dose of the vaccine, when administered to infants in a three-dose schedule at 6, 10 and 14 weeks of age.

The study will also assess the reactogenicity of the vaccine 7 days after each vaccination and safety from first vaccination up to 4 weeks after the last vaccination with ROTAVAC® and ROTAVAC 5D, and of Rotarix® when administered to infants in a two-dose schedule at 6 and 10 weeks of age.

DETAILED DESCRIPTION:
This study is designed as a Phase IIb, single center, randomized, controlled, open label study with 3 groups of infants (n=150 per group) receiving either three doses of ROTAVAC® three doses of ROTAVAC 5D or two doses of Rotarix®. 450 participants will be randomized (1:1:1) to receive ROTAVAC®, ROTAVAC 5D or Rotarix®. The three doses of ROTAVAC® and ROTAVAC 5D will be administered at 6, 10 and 14 weeks of age whereas two doses of Rotarix® will be administered at 6 and 10 weeks of age. All vaccines will be administered concomitantly with EPI vaccines including Diphtheria, Tetanus, Pertussis, Haemophilus influenzae type b and Hepatitis B vaccine (DTwP-Hib-HepB), Pneumococcal conjugate vaccine and OPV at 6, 10 and 14 weeks and IPV at week 14 (when switched to in Zambia). The participants will be monitored for 30 minutes following vaccine administration for immediate adverse events.

A blood sample will be obtained from all the participating infants before first vaccination and four weeks after the last vaccine dose. This would mean that the blood sample will be collected at approximately 14 weeks of age for infants in the Rotarix® arm and 18 weeks for infants in the ROTAVAC® groups.

Enhanced passive/Active surveillance for vaccine reactogenicity (solicited reactions) over the 7-day period after each vaccination will be conducted on all infants. In addition, surveillance for unsolicited AEs, SAEs including intussusception will be carried out over the period between first vaccination and four weeks after the last vaccination on all infants.

The study will compare the immunogenicity of the two formulations of ROTAVAC® i.e. ROTAVAC® vs. ROTAVAC 5D and will descriptively analyze the immune response to Rotarix®. Primary immunogenicity analysis of all samples will be based on a validated ELISA which uses strain WC3 as a substrate. A subset of the samples (50 pairs/arms) collected will also be tested by a validated ELISA which uses strain 89-12 (G1P8 virus) as a substrate. This trial will generate immunogenicity and safety data on ROTAVAC® and ROTAVAC 5D outside of India. Presentation of data to Zambian Ministry of Health, WHO and in peer reviewed open access publications will be key audiences targeted for communication of results.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infant as established by medical history and clinical examination before entering the study.
2. Age: 6-8 weeks (42-56 days, both days inclusive) confirmed by Immunization Record.
3. Infants received age-appropriate EPI vaccines till enrolment.
4. Ability and willingness to provide informed consent as per local consenting procedures.
5. Parent can be contacted on phone and confirms intention to remain in the study area with the participant during the study period.

Exclusion Criteria:

1. Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrolment (temporary exclusion).
2. Presence of fever on the day of enrolment (temporary exclusion).
3. Acute disease at the time of enrolment (temporary exclusion).
4. Concurrent participation in another clinical trial throughout the entire timeframe of this study.
5. Presence of severe malnutrition (weight-for-height z-score < -3SD median).
6. Any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would compromise the child's health or is likely to result in non-conformance to the protocol.
7. History of congenital abdominal disorders, intussusception, abdominal surgery
8. Known or suspected impairment of immunological function based on medical history and physical examination.
9. Prior receipt or intent to receive rotavirus and other age specified EPI vaccines outside of the study center and during study participation.
10. A known sensitivity or allergy to any component of the study vaccine.
11. Clinically detectable significant congenital or genetic defect.
12. History of persistent diarrhea (defined as diarrhea more than 14 days).
13. Participant's parents not able, available or willing to accept active follow-up by the study staff.
14. Has received any immunoglobulin therapy and/or blood products since birth or planned administration during the study period.
15. History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study.
16. History of any neurologic disorders or seizures.
17. Any medical condition in the parents/infants that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parent's/legally acceptable representative's ability to give informed consent.
18. Participant is a direct descendant (child or grandchild) of any person employed by the Sponsor, the CRO, the PI or study site personnel.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Rathi, MD, Study Director — PATH
Locations (1):
- George Research Centre, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tate JE, Burton AH, Boschi-Pinto C, Parashar UD; World Health Organization-Coordinated Global Rotavirus Surveillance Network. Global, Regional, and National Estimates of Rotavirus Mortality in Children <5 Years of Age, 2000-2013. Clin Infect Dis. 2016 May 1;62 Suppl 2(Suppl 2):S96-S105. doi: 10.1093/cid/civ1013. PMID 27059362
- [Background] Atherly DE, Lewis KD, Tate J, Parashar UD, Rheingans RD. Projected health and economic impact of rotavirus vaccination in GAVI-eligible countries: 2011-2030. Vaccine. 2012 Apr 27;30 Suppl 1(Suppl 1):A7-14. doi: 10.1016/j.vaccine.2011.12.096. PMID 22520139
- [Background] Beres LK, Tate JE, Njobvu L, Chibwe B, Rudd C, Guffey MB, Stringer JS, Parashar UD, Chilengi R. A Preliminary Assessment of Rotavirus Vaccine Effectiveness in Zambia. Clin Infect Dis. 2016 May 1;62 Suppl 2(Suppl 2):S175-82. doi: 10.1093/cid/civ1206. PMID 27059353
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Chilengi R, Simuyandi M, Beach L, Mwila K, Becker-Dreps S, Emperador DM, Velasquez DE, Bosomprah S, Jiang B. Association of Maternal Immunity with Rotavirus Vaccine Immunogenicity in Zambian Infants. PLoS One. 2016 Mar 14;11(3):e0150100. doi: 10.1371/journal.pone.0150100. eCollection 2016. PMID 26974432
- [Background] Tate JE, Yen C, Steiner CA, Cortese MM, Parashar UD. Intussusception Rates Before and After the Introduction of Rotavirus Vaccine. Pediatrics. 2016 Sep;138(3):e20161082. doi: 10.1542/peds.2016-1082. Epub 2016 Aug 24. PMID 27558938
- [Background] Madhi SA, Cunliffe NA, Steele D, Witte D, Kirsten M, Louw C, Ngwira B, Victor JC, Gillard PH, Cheuvart BB, Han HH, Neuzil KM. Effect of human rotavirus vaccine on severe diarrhea in African infants. N Engl J Med. 2010 Jan 28;362(4):289-98. doi: 10.1056/NEJMoa0904797. PMID 20107214
- [Background] Armah GE, Sow SO, Breiman RF, Dallas MJ, Tapia MD, Feikin DR, Binka FN, Steele AD, Laserson KF, Ansah NA, Levine MM, Lewis K, Coia ML, Attah-Poku M, Ojwando J, Rivers SB, Victor JC, Nyambane G, Hodgson A, Schodel F, Ciarlet M, Neuzil KM. Efficacy of pentavalent rotavirus vaccine against severe rotavirus gastroenteritis in infants in developing countries in sub-Saharan Africa: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Aug 21;376(9741):606-14. doi: 10.1016/S0140-6736(10)60889-6. Epub 2010 Aug 6. PMID 20692030
- [Background] Zaman K, Dang DA, Victor JC, Shin S, Yunus M, Dallas MJ, Podder G, Vu DT, Le TP, Luby SP, Le HT, Coia ML, Lewis K, Rivers SB, Sack DA, Schodel F, Steele AD, Neuzil KM, Ciarlet M. Efficacy of pentavalent rotavirus vaccine against severe rotavirus gastroenteritis in infants in developing countries in Asia: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Aug 21;376(9741):615-23. doi: 10.1016/S0140-6736(10)60755-6. Epub 2010 Aug 6. PMID 20692031
- [Background] Bhandari N, Rongsen-Chandola T, Bavdekar A, John J, Antony K, Taneja S, Goyal N, Kawade A, Kang G, Rathore SS, Juvekar S, Muliyil J, Arya A, Shaikh H, Abraham V, Vrati S, Proschan M, Kohberger R, Thiry G, Glass R, Greenberg HB, Curlin G, Mohan K, Harshavardhan GV, Prasad S, Rao TS, Boslego J, Bhan MK; India Rotavirus Vaccine Group. Efficacy of a monovalent human-bovine (116E) rotavirus vaccine in Indian infants: a randomised, double-blind, placebo-controlled trial. Lancet. 2014 Jun 21;383(9935):2136-43. doi: 10.1016/S0140-6736(13)62630-6. Epub 2014 Mar 12. PMID 24629994
- [Background] Isanaka S, Guindo O, Langendorf C, Matar Seck A, Plikaytis BD, Sayinzoga-Makombe N, McNeal MM, Meyer N, Adehossi E, Djibo A, Jochum B, Grais RF. Efficacy of a Low-Cost, Heat-Stable Oral Rotavirus Vaccine in Niger. N Engl J Med. 2017 Mar 23;376(12):1121-1130. doi: 10.1056/NEJMoa1609462. PMID 28328346
- [Background] Mpabalwani EM, Simwaka CJ, Mwenda JM, Mubanga CP, Monze M, Matapo B, Parashar UD, Tate JE. Impact of Rotavirus Vaccination on Diarrheal Hospitalizations in Children Aged <5 Years in Lusaka, Zambia. Clin Infect Dis. 2016 May 1;62 Suppl 2(Suppl 2):S183-7. doi: 10.1093/cid/civ1027. PMID 27059354
- [Background] Bishop R. Discovery of rotavirus: Implications for child health. J Gastroenterol Hepatol. 2009 Oct;24 Suppl 3:S81-5. doi: 10.1111/j.1440-1746.2009.06076.x. PMID 19799704
- [Background] Santos N, Hoshino Y. Global distribution of rotavirus serotypes/genotypes and its implication for the development and implementation of an effective rotavirus vaccine. Rev Med Virol. 2005 Jan-Feb;15(1):29-56. doi: 10.1002/rmv.448. PMID 15484186
- [Background] Kang G, Arora R, Chitambar SD, Deshpande J, Gupte MD, Kulkarni M, Naik TN, Mukherji D, Venkatasubramaniam S, Gentsch JR, Glass RI, Parashar UD; Indian Rotavirus Strain Surveillance Network. Multicenter, hospital-based surveillance of rotavirus disease and strains among indian children aged <5 years. J Infect Dis. 2009 Nov 1;200 Suppl 1:S147-53. doi: 10.1086/605031. PMID 19817593
- [Background] Rodrigo C, Salman N, Tatochenko V, Meszner Z, Giaquinto C. Recommendations for rotavirus vaccination: A worldwide perspective. Vaccine. 2010 Jul 12;28(31):5100-8. doi: 10.1016/j.vaccine.2010.04.108. Epub 2010 May 14. PMID 20472032
- [Background] Simpson E, Wittet S, Bonilla J, Gamazina K, Cooley L, Winkler JL. Use of formative research in developing a knowledge translation approach to rotavirus vaccine introduction in developing countries. BMC Public Health. 2007 Oct 5;7:281. doi: 10.1186/1471-2458-7-281. PMID 17919334
- [Background] Levy K, Hubbard AE, Eisenberg JN. Seasonality of rotavirus disease in the tropics: a systematic review and meta-analysis. Int J Epidemiol. 2009 Dec;38(6):1487-96. doi: 10.1093/ije/dyn260. Epub 2008 Dec 4. PMID 19056806
- [Background] Atchison CJ, Tam CC, Hajat S, van Pelt W, Cowden JM, Lopman BA. Temperature-dependent transmission of rotavirus in Great Britain and The Netherlands. Proc Biol Sci. 2010 Mar 22;277(1683):933-42. doi: 10.1098/rspb.2009.1755. Epub 2009 Nov 25. PMID 19939844
- [Background] Ruiz-Palacios GM, Perez-Schael I, Velazquez FR, Abate H, Breuer T, Clemens SC, Cheuvart B, Espinoza F, Gillard P, Innis BL, Cervantes Y, Linhares AC, Lopez P, Macias-Parra M, Ortega-Barria E, Richardson V, Rivera-Medina DM, Rivera L, Salinas B, Pavia-Ruz N, Salmeron J, Ruttimann R, Tinoco JC, Rubio P, Nunez E, Guerrero ML, Yarzabal JP, Damaso S, Tornieporth N, Saez-Llorens X, Vergara RF, Vesikari T, Bouckenooghe A, Clemens R, De Vos B, O'Ryan M; Human Rotavirus Vaccine Study Group. Safety and efficacy of an attenuated vaccine against severe rotavirus gastroenteritis. N Engl J Med. 2006 Jan 5;354(1):11-22. doi: 10.1056/NEJMoa052434. PMID 16394298
- [Background] Bhandari N, Rongsen-Chandola T, Bavdekar A, John J, Antony K, Taneja S, Goyal N, Kawade A, Kang G, Rathore SS, Juvekar S, Muliyil J, Arya A, Shaikh H, Abraham V, Vrati S, Proschan M, Kohberger R, Thiry G, Glass R, Greenberg HB, Curlin G, Mohan K, Harshavardhan GV, Prasad S, Rao TS, Boslego J, Bhan MK; India Rotavirus Vaccine Group. Efficacy of a monovalent human-bovine (116E) rotavirus vaccine in Indian children in the second year of life. Vaccine. 2014 Aug 11;32 Suppl 1:A110-6. doi: 10.1016/j.vaccine.2014.04.079. PMID 25091663
- [Background] Ward RL, Bernstein DI. Protection against rotavirus disease after natural rotavirus infection. US Rotavirus Vaccine Efficacy Group. J Infect Dis. 1994 Apr;169(4):900-4. doi: 10.1093/infdis/169.4.900. PMID 8133107
- [Background] Bhan MK, Lew JF, Sazawal S, Das BK, Gentsch JR, Glass RI. Protection conferred by neonatal rotavirus infection against subsequent rotavirus diarrhea. J Infect Dis. 1993 Aug;168(2):282-7. doi: 10.1093/infdis/168.2.282. PMID 8393054
- [Background] Aiyar J, Bhan MK, Bhandari N, Kumar R, Raj P, Sazawal S. Rotavirus-specific antibody response in saliva of infants with rotavirus diarrhea. J Infect Dis. 1990 Dec;162(6):1383-4. doi: 10.1093/infdis/162.6.1383. PMID 2172405
- [Background] Appaiahgari MB, Glass R, Singh S, Taneja S, Rongsen-Chandola T, Bhandari N, Mishra S, Vrati S. Transplacental rotavirus IgG interferes with immune response to live oral rotavirus vaccine ORV-116E in Indian infants. Vaccine. 2014 Feb 3;32(6):651-6. doi: 10.1016/j.vaccine.2013.12.017. Epub 2013 Dec 25. PMID 24374502
- [Background] Bishop RF, Barnes GL, Cipriani E, Lund JS. Clinical immunity after neonatal rotavirus infection. A prospective longitudinal study in young children. N Engl J Med. 1983 Jul 14;309(2):72-6. doi: 10.1056/NEJM198307143090203. PMID 6304516
- [Background] Glass RI, Bhan MK, Ray P, Bahl R, Parashar UD, Greenberg H, Rao CD, Bhandari N, Maldonado Y, Ward RL, Bernstein DI, Gentsch JR. Development of candidate rotavirus vaccines derived from neonatal strains in India. J Infect Dis. 2005 Sep 1;192 Suppl 1:S30-5. doi: 10.1086/431498. PMID 16088802
- [Background] Ing DJ, Glass RI, Woods PA, Simonetti M, Pallansch MA, Wilcox WD, Davidson BL, Sievert AJ. Immunogenicity of tetravalent rhesus rotavirus vaccine administered with buffer and oral polio vaccine. Am J Dis Child. 1991 Aug;145(8):892-7. doi: 10.1001/archpedi.1991.02160080070023. PMID 1650128
- [Background] Clark HF, Burke CJ, Volkin DB, Offit P, Ward RL, Bresee JS, Dennehy P, Gooch WM, Malacaman E, Matson D, Walter E, Watson B, Krah DL, Dallas MJ, Schodel F, Kaplan kM, Heaton P. Safety, immunogenicity and efficacy in healthy infants of G1 and G2 human reassortant rotavirus vaccine in a new stabilizer/buffer liquid formulation. Pediatr Infect Dis J. 2003 Oct;22(10):914-20. doi: 10.1097/01.inf.0000091887.48999.77. PMID 14551493
- [Background] Kerdpanich A, Chokephaibulkit K, Watanaveeradej V, Vanprapar N, Simasathien S, Phavichitr N, Bock HL, Damaso S, Hutagalung Y, Han HH. Immunogenicity of a live-attenuated human rotavirus RIX4414 vaccine with or without buffering agent. Hum Vaccin. 2010 Mar 26;6(3):10428. doi: 10.4161/hv.6.3.10428. Epub 2010 Mar 26. PMID 20220306
- [Background] Estes MK, Graham DY, Smith EM, Gerba CP. Rotavirus stability and inactivation. J Gen Virol. 1979 May;43(2):403-9. doi: 10.1099/0022-1317-43-2-403. PMID 39115
- [Background] Weiss C, Clark HF. Rapid inactivation of rotaviruses by exposure to acid buffer or acidic gastric juice. J Gen Virol. 1985 Dec;66 ( Pt 12):2725-30. doi: 10.1099/0022-1317-66-12-2725. PMID 2999315
- [Background] Feng N, Burns JW, Bracy L, Greenberg HB. Comparison of mucosal and systemic humoral immune responses and subsequent protection in mice orally inoculated with a homologous or a heterologous rotavirus. J Virol. 1994 Dec;68(12):7766-73. doi: 10.1128/JVI.68.12.7766-7773.1994. PMID 7966566
- [Background] Graham DY, Dufour GR, Estes MK. Minimal infective dose of rotavirus. Arch Virol. 1987;92(3-4):261-71. doi: 10.1007/BF01317483. PMID 3028333
- [Background] Ward RL, Kirkwood CD, Sander DS, Smith VE, Shao M, Bean JA, Sack DA, Bernstein DI. Reductions in cross-neutralizing antibody responses in infants after attenuation of the human rotavirus vaccine candidate 89-12. J Infect Dis. 2006 Dec 15;194(12):1729-36. doi: 10.1086/509623. Epub 2006 Nov 6. PMID 17109346
- [Background] Mandomando I, Weldegebriel G, de Deus N, Mwenda JM. Feasibility of using regional sentinel surveillance to monitor the rotavirus vaccine impact, effectiveness and intussusception incidence in the African Region. Vaccine. 2017 Mar 23;35(13):1663-1667. doi: 10.1016/j.vaccine.2017.01.072. Epub 2017 Mar 1. PMID 28242070
- [Background] Bhandari N, Sharma P, Glass RI, Ray P, Greenberg H, Taneja S, Saksena M, Rao CD, Gentsch JR, Parashar U, Maldonado Y, Ward RL, Bhan MK. Safety and immunogenicity of two live attenuated human rotavirus vaccine candidates, 116E and I321, in infants: results of a randomised controlled trial. Vaccine. 2006 Jul 26;24(31-32):5817-23. doi: 10.1016/j.vaccine.2006.05.001. Epub 2006 May 12. PMID 16735085
- [Background] Bhandari N, Sharma P, Taneja S, Kumar T, Rongsen-Chandola T, Appaiahgari MB, Mishra A, Singh S, Vrati S; Rotavirus Vaccine Development Group. A dose-escalation safety and immunogenicity study of live attenuated oral rotavirus vaccine 116E in infants: a randomized, double-blind, placebo-controlled trial. J Infect Dis. 2009 Aug 1;200(3):421-9. doi: 10.1086/600104. PMID 19545211
- [Background] Chandola TR, Taneja S, Goyal N, Antony K, Bhatia K, More D, Bhandari N, Cho I, Mohan K, Prasad S, Harshavardhan G, Rao TS, Vrati S, Bhan MK. ROTAVAC(R) does not interfere with the immune response to childhood vaccines in Indian infants: A randomized placebo controlled trial. Heliyon. 2017 May 16;3(5):e00302. doi: 10.1016/j.heliyon.2017.e00302. eCollection 2017 May. PMID 28560356
- [Background] Ella R, Bobba R, Muralidhar S, Babji S, Vadrevu KM, Bhan MK. A Phase 4, multicentre, randomized, single-blind clinical trial to evaluate the immunogenicity of the live, attenuated, oral rotavirus vaccine (116E), ROTAVAC(R), administered simultaneously with or without the buffering agent in healthy infants in India. Hum Vaccin Immunother. 2018 Jul 3;14(7):1791-1799. doi: 10.1080/21645515.2018.1450709. Epub 2018 Apr 12. PMID 29543547
- See also: Rotarix (Product Information). — https://www.gsksource.com/pharma/content/dam/GlaxoSmithKline/US/en/Prescribing_Information/Rotarix/pdf/ROTARIX-PI-PIL.PDF
- See also: Rotateq (Product Information). — https://www.merck.com/product/usa/pi_circulars/r/rotateq/rotateq_ppi.pdf
- See also: PATH welcomes new promising study results for rotavirus vaccine candidate. — https://www.path.org/media-center/path-welcomes-new-promising-study-results-for-rotavirus-vaccine-candidate/
- See also: Bharat Biotech receives National Technology Award for Rotavac from President of India — http://www.pharmabiz.com/NewsDetails.aspx?aid=108851&sid=2

RESULTS

PARTICIPANT FLOW:
Groups:
- ROTAVAC 5D®: ROTAVAC 5D® administered at 6, 10 and 14 weeks of age.
- ROTAVAC®: ROTAVAC® administered at 6, 10 and 14 weeks of age.
- Rotarix®: Rotarix® administered at 6 and 10 weeks of age.
Period: Overall Study
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Started | 150 | 150 | 150
Completed | 131 | 132 | 139
Not Completed | 19 | 18 | 11
Not completed — Withdrawal by Subject | 7 | 9 | 7
Not completed — Lost to Follow-up | 5 | 6 | 0
Not completed — Protocol Violation | 3 | 0 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — migration | 2 | 3 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix® | Total
Number analyzed (Participants) | 150 | 150 | 150 | 450
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 6.56 (0.477) | 6.50 (0.473) | 6.60 (0.491) | 6.55 (0.475)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 77 | 66 | 209
  Male | 84 | 73 | 84 | 241
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 150 | 150 | 150 | 450
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Zambia | 150 | 150 | 150 | 450

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration Using WC3 as the Viral Lysate
Description: GMC of serum anti-rotavirus IgA antibodies as measured by enzyme linked immunosorbent assay (ELISA) using WC3 (heterologous to vaccine strain) as the viral lysate. WC3 strain of rotavirus used in the ELISA assay was heterologous to the 116E strain contained in the vaccines ROTAVAC 5D® and ROTAVAC®.
Time Frame: 28 day after last dose of the study vaccine
Population: The analysis was performed on Per Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: U/ml
Arm/Group | ROTAVAC 5D® | ROTAVAC®
Number analyzed (Participants) | 128 | 124
U/ml | 18.1 [13.7 to 24.0] | 14.0 [10.4 to 18.8]
Statistical Analysis 1: Comparison: ROTAVAC 5D® vs ROTAVAC®; Test type: Non-Inferiority — If the lower limit of the 95% CI of the ratio of GMCs between the ROTAVAC 5D® and ROTAVAC® groups was larger than 1/2 (i.e. > 0.5), ROTAVAC 5D® would be considered non-inferior to ROTAVAC®; t-test, 2 sided; GMC ratio = 1.294, 95% CI 2-sided [0.862 to 1.924]

2. Secondary Outcome: Immediate Adverse Events
Description: Percentage of participants reporting immediate adverse events after each vaccination
Time Frame: within 30 minutes' post-vaccination.
Population: The analysis was performed on Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- ROTAVAC®: ROTAVAC ® administered at 6, 10 and 14 weeks of age.
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 150 | 150 | 150
Participants | 1 | 0 | 1

3. Secondary Outcome: Solicited Adverse Events
Description: Percentage of participants reporting solicited post-vaccination reactogenicity (fever, diarrhea, vomiting, decreased appetite, irritability, decreased activity level)
Time Frame: 7 day period after each vaccination.
Population: The analysis was performed on Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 146 | 144 | 146
Participants
  Any Solicited AEs | 138 | 136 | 129
  Fever | 110 | 109 | 100
  Diarrhea | 15 | 11 | 8
  Vomiting | 14 | 14 | 15
  Decreased appetite | 53 | 44 | 44
  Decreased activity level | 62 | 66 | 55
  Irritability | 105 | 109 | 101

4. Secondary Outcome: Unsolicited Adverse Events
Description: Percentage of participants reporting unsolicited AEs at a rate >5%.
Time Frame: From first vaccination through 4 weeks after the last vaccination.
Population: The analysis was performed on Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 137 | 139 | 142
Participants
  Any Unsolicited AEs | 93 | 95 | 81
  Conjunctivitis | 10 | 10 | 6
  Rhinitis | 21 | 12 | 10
  Upper respiratory tract infection | 52 | 46 | 39
  Diarrhoea | 18 | 17 | 11

5. Secondary Outcome: Serious Adverse Events
Description: Percentage of participants reporting SAEs
Time Frame: From first vaccination through 4 weeks after the last vaccination of each study participant. Immunogenicity
Population: The analysis was performed on Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 137 | 139 | 142
Participants
  Any SAEs | 2 | 1 | 3
  Diarrhoea | 1 | 0 | 0
  Bronchiolitis | 1 | 0 | 2
  Sepsis | 0 | 1 | 1

6. Secondary Outcome: Seroconversion Rate in Each of the Three Arms as Measured by ELISA Using WC3 as the Viral Lysate
Description: Seroconversion is defined as a post-vaccination serum anti-rotavirus IgA antibody concentration of at least 20 U/mL if a baseline concentration is < 20 U/mL or a post-vaccination serum anti-rotavirus IgA antibody concentration of ≥ 2-fold baseline level if a baseline concentration is ≥ 20 U/mL.
  WC3 strain of rotavirus used in the ELISA assay was heterologous to the 116E strain contained in the vaccines ROTAVAC® and ROTAVAC 5D®.
Time Frame: 28 days after last dose of study vaccine.
Population: The analysis was performed on Per Protocol Population
Measure: Count of Participants; unit: Participants
Groups:
- Rotarix®: Rotarix® administered at6 and 10 weeks of age
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 128 | 124 | 136
Participants | 52 | 41 | 50

7. Secondary Outcome: Seropositivity Rate in Each of the Three Vaccine Arms as Measured by ELISA Using WC3 as the Viral Lysate
Description: Seropositivity is defined as serum anti-rotavirus IgA antibody concentration ≥ 20 U/mL. WC3 strain of rotavirus used in the ELISA assay was heterologous to the 116E strain contained in the vaccines ROTAVAC® and ROTAVAC 5D®.
Time Frame: 28 days after last dose of study vaccine
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 128 | 124 | 136
Participants | 54 | 42 | 52

8. Secondary Outcome: Seroresponse Rate in Each of the Three Vaccine Arms as Measured by ELISA Using WC3 as the Viral Lysate
Description: Seroresponse will be assessed as a four-fold, three-fold and two- fold rise in antibody concentration from baseline. Seroresponse will be assessed as a four-fold, three-fold and two-fold rise in antibody concentration from baseline. WC3 strain of rotavirus used in the ELISA assay was heterologous to the 116E strain contained in the vaccines ROTAVAC® and ROTAVAC 5D®.
Time Frame: 28 days after last dose of study vaccine
Population: The analysis was performed on Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 128 | 124 | 136
Participants
  Seroresponse rate- Two-fold rise | 79 | 65 | 74
  Seroresponse rate- Three-fold rise | 71 | 55 | 66
  Seroresponse rate- Four-fold rise | 61 | 49 | 58

9. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Each of the Three Vaccine Arms as Measured by ELISA Using WC3 as the Viral Lysate
Description: GMFR in each of the ROTAVAC 5D®, ROTAVAC® and Rotarix® vaccine arms. WC3 strain of rotavirus used in the ELISA assay was heterologous to the 116E strain contained in the vaccines ROTAVAC® and ROTAVAC 5D®.
Time Frame: At 28 days after last dose of study vaccine in reference to baseline.
Population: The analysis was performed on Per Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 128 | 124 | 136
Fold rise | 4.6 [3.5 to 6.1] | 3.6 [2.7 to 4.9] | 3.8 [2.9 to 4.9]

10. Other Pre Specified Outcome: Geometric Mean Concentrations Using Strain 89-12 as the Viral Lysate
Description: GMCs of serum anti-rotavirus IgA antibodies in each of the three vaccine arms. 89-12 strain of Rotavirus used in the ELISA assay was homologous to Rotarix® and was heterologous to the strain contained in ROTAVAC® and ROTAVAC 5D®.
Time Frame: 28 days after the last dose of a study vaccine.
Population: The analysis was performed on Per Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: Au/ml
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 50 | 50 | 50
Au/ml | 20.6 [12.4 to 34.1] | 19.2 [11.0 to 33.5] | 38.0 [20.5 to 70.6]

11. Other Pre Specified Outcome: Seroconversion Using Strain 89-12 as the Viral Lysate
Description: Seroconversion rate in three vaccine arms. 89-12 strain of Rotavirus used in the ELISA assay was homologous to Rotarix® and was heterologous to the strain contained in ROTAVAC® and ROTAVAC 5D®.
Time Frame: 28 days after the last dose of a study vaccine.
Population: The analysis was performed on Per Protocol Population
Measure: Count of Participants; unit: Participants
Groups:
- ROTAVAC 5D®: ROTAVAC 5D® administered at 6,10 and14 weeks of age.
- ROTAVAC®: ROTAVAC® administered at 6,10 and14 weeks of age.
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 50 | 50 | 50
Participants | 24 | 18 | 26

12. Other Pre Specified Outcome: Seropositivity Using Strain 89-12 as the Viral Lysate
Description: Seropositivity rate in three vaccine arms. 89-12 strain of Rotavirus used in the ELISA assay was homologous to Rotarix® and was heterologous to the strain contained in ROTAVAC® and ROTAVAC 5D®.
Time Frame: at baseline and 28 days after last dose of study vaccine
Population: The analysis was performed on Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 50 | 50 | 50
Participants | 25 | 18 | 27

13. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) Using Strain 89-12 as the Viral Lysate
Description: GMFR in the three vaccine arms. 89-12 strain of Rotavirus used in the ELISA assay was homologous to Rotarix® and was heterologous to the strain contained in ROTAVAC® and ROTAVAC 5D®.
Time Frame: at 28 days after last dose of study vaccine in reference to baseline.
Population: The analysis was performed on Per Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
Number analyzed (Participants) | 50 | 50 | 50
Fold rise | 4.8 [3.0 to 7.8] | 4.9 [2.8 to 8.7] | 8.8 [4.7 to 16.4]

ADVERSE EVENTS:
Time Frame: Immediate Adverse Event within 30 mins post vaccination. Solicited adverse events for 7 days post vaccination. Unsolicited Adverse events for 28 days after each vaccination. Serious Adverse Events.
Arm/Group | ROTAVAC 5D® | ROTAVAC® | Rotarix®
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 2/137 | 1/139 | 3/142
Other Adverse Events (participants affected / at risk) | 93/137 | 95/139 | 81/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ROTAVAC 5D® (N=137) | ROTAVAC® (N=139) | Rotarix® (N=142)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ROTAVAC 5D® (N=137) | ROTAVAC® (N=139) | Rotarix® (N=142)
Conjuntivities (Infections and infestations) | 10 (10) | 10 (10) | 6 (6)
Rhinitis (Infections and infestations) | 21 (22) | 12 (12) | 10 (10)
Respiratory Tract Infection (Infections and infestations) | 22 (23) | 26 (27) | 15 (16)
Upper Respiratory Tract Infection (Infections and infestations) | 52 (71) | 46 (56) | 39 (43)
Diarrhoea (Infections and infestations) | 18 (18) | 17 (18) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03602053/SAP_000.pdf
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03602053/Prot_001.pdf